CLINICAL TRIAL: NCT06811363
Title: Contribution of Bone to Urine Citrate
Status: Not yet recruiting | Type: Observational
Sponsor: University of Texas Southwestern Medical Center (Other)
Responsible Party: Principal Investigator, Eleanor Lederer, Professor, University of Texas Southwestern Medical Center
Other Study IDs: STU-2024-0760
Record Dates: First submitted 2025-01-31; First posted 2025-02-06 (Actual); Last update posted 2025-12-22 (Actual); Status verified 2025-08

CONDITIONS: Osteoporosis
Keywords: naïve to treatment; bone mass; bone turnover
MeSH Terms: conditions — Osteoporosis | interventions — Metabolic Networks and Pathways; Anabolic Agents

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Anti-resorptive agents use Group: Patients with osteoporosis naïve to treatment will initiate treatment with anti-resorptive agents (zoledronic acid or denosumab)
  Interventions: Other: Metabolic / prescribed diet; Other: KCit Load (40 meq); Drug: Anti-resorptive agents
- Anabolic agents use Group: Patients with osteoporosis naïve to treatment will initiate treatment with anabolic agents (romosozumab)
  Interventions: Other: Metabolic / prescribed diet; Other: KCit Load (40 meq); Drug: Anabolic Agents

INTERVENTIONS:
Other: Metabolic / prescribed diet — Instructed diet (400 mg Ca, 800 mg P, 100 mEq Na) and two liters of distilled water daily for three days (equilibration period), followed by a constant standardized meal with the same composition of Ca, P, and Na for one day. After 240hr urine sample collection patient fasted the preceding evening except for 300 ml of distilled water at 9 pm and 11 pm. On test days, 600 ml distilled water given and fasting blood obtained.
Other: KCit Load (40 meq) — Potassium citrate load of 40meq will be given after fasting blood has been obtained
Drug: Anti-resorptive agents — Zoledronic acid or Denosumab (as prescribed by their physician)
  Groups: Anti-resorptive agents use Group
Drug: Anabolic Agents — Romosozumab (as prescribed by their physician)
  Groups: Anabolic agents use Group

SUMMARY:
Identification of the mechanisms by which bone contributes to urine citrate could lead to alternative explanations for and approaches to hypocitraturia. This proposal to explore the role of bone in urine citrate addresses the mission of the CMMCR to discover new mechanisms and innovative therapies for diseases of mineral metabolism. The results will be used to apply for extramural funding to further examine the nonrenal regulation of UCit.

Hypothesis: Serum citrate is a function of bone citrate formation dependent on both bone mass and bone turnover. 20 subjects with osteoporosis naïve to treatment will be identified to examine bone parameters that correlate with ΔUcit/Δk.

Use of potent anti-osteoporotic therapies to increase the likelihood of identifying significant bone turnover and BMD correlations with ΔUcit/Uk will take place in this study.

Plan to achieve the following aim:

* Correlate ∆ Ucit/∆k in response to acute KCit load with:

  1. Bone turnover marker at baseline
  2. BMD at baseline
  3. Change in bone turnover markers at 1 month and 6 months with each osteoporosis treatment modality (anti-resorptive agents such as Zoledronic acid or Denosumab, or the Anabolic agent Romosozumab)
  4. Change in bone mineral density at 6 with each osteoporosis treatment modality (anti-resorptive agents such as Zoledronic acid or Denosumab, or the Anabolic agent Romosozumab)

DETAILED DESCRIPTION:
Screening Visit: Before enrollment into the trial, potential candidates will undergo screening, whereby the study team will conduct a physical exam and ask questions about the subject's medical history, including medications and any surgical procedures. Those who meet the entry-exclusion criteria will be selected for consideration into the study. During screening, subjects will provide information on or have the following exams, tests or procedures:

* Social and medical history;
* Medications;
* Vital signs;
* Demographic information (age, gender, ethnic origin);
* Personal information (name, date of birth, address, telephone number, emergency contact, and referring physician)

Assignment to groups:

Group 1- Patients with osteoporosis naïve to treatment will initiate treatment with anti-resorptive agents (zoledronic acid or denosumab).

Group 2- - Patients with osteoporosis naïve to treatment will initiate treatment with anabolic agents (romosozumab).

The anti-osteoporosis medication would be prescribed by the treating physician.

Phase 1 (pre-treatment phase):

All patients will be stabilized with instructed diet (400 mg Ca, 800 mg P, 100 mEq Na) and two liters of distilled water daily for three days (equilibration period), followed by a constant standardized meal with the same composition of Ca, P, and Na for one day (stabilization period) and undergo a run-in (pre-Rx) period.

One 24-hour urine will be obtained on day 4 without mineral oil (stabilization period). The 24-hour urine will be analyzed for total volume, pH, creatinine, sodium, potassium, calcium, magnesium, phosphorus chloride, oxalate, citrate, ammonium, titratable acidity, bicarbonate and deoxypyridinoline (DPD). The patient will be fasted from 9 pm of the preceding evening except for 300 ml of distilled water at 9 pm and 11 pm. On test days, 600 ml of distilled water will be given at 7 am and fasting blood will be obtained tested for Serum BMP, citrate and bone turnover markers (CTX, P1NP, bone alkaline phosphatase).

Potassium citrate load of 40meq will be given after fasting blood has been obtained and hourly blood and urine measurements of citrate and creatinine for 4 hours after ingesting will be collected.

Laboratory Analysis:

Urine samples - Post-load every 1 hour for 4 hours analyzed for citrate and creatinine by Mineral Metabolism Laboratory.

Blood samples - Post-load every 1 hour for 4 hours analyzed for citrate and creatinine by Mineral Metabolism Laboratory.

Phase 2 (1 month after initiating treatment) and Phase 3 (6 months after initiating treatment):

These two visits consist of identical study procedure as Phase 1.

Imaging:

Imagining studies will be done using DXA for bone density measurement and micro-CT measurement for determaination of bone quality and microarchitecture of the bone. The imaging studies will be performed during phase 1 and phase 3.

ELIGIBILITY:
Inclusion Criteria:

* Osteoporosis naïve to treatment

Exclusion Criteria:

* eGFR < 60 ml/min
* chronic diarrhea or gastrointestinal illness

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with osteoporosis
Sampling Method: Non-Probability Sample
Enrollment: 25 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2026-03 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Correlation of change in Urine Citrate levels to change in Potassium levels with change in bone turnover markers at 1 month after initiating treatment | Baseline, 1month after initiating treatment
  Change in Urine Citrate levels to change in Potassium levels from the 24h urine samples is measured and will be correlated with baseline and post treatment bone turnover markers by multiple linear regression modeling using forward and backward selection.
Correlation of change in Urine Citrate levels to change in Potassium levels with change in bone turnover markers at 6 months after initiating treatment | Baseline, 6 months after initiating treatment
  Change in Urine Citrate levels to change in Potassium levels from the 24h urine samples is measured and will be correlated with baseline and post treatment bone turnover markers by multiple linear regression modeling using forward and backward selection.
Correlation of change in Urine Citrate levels to change in Potassium levels with bone densitometry at baseline | Baseline
  Change in Urine Citrate levels to change in Potassium levels will be correlated with bone densitometry at lumbar spine, right hip, and radius
Correlation of change in Urine Citrate levels to change in Potassium levels with change in bone densitometry at 6 months after initiating treatment | Baseline, 6 months after initiating treatment
  Change in Urine Citrate levels to change in Potassium levels will be correlated with change in bone densitometry at lumbar spine, right hip, and radius
K Cit load | Predose, 0.5, 1, 2, 3, 4 hours after drug administration in Phases 1, 2, 3
  The AUC for citrate will be calculated from the serum and urine levels based on the assumption that oral K Cit is 100% absorbed to estimate hepatic uptake effect on filtered load. The fractional excretion of citrate (FeCit) will be calculated from hourly serum and urine creatinine and citrate levels (FeCit = (serum Cit x Urine Cr)/urine Cit x serum Cr) x 100. Differences in FeCit will be correlated with ΔUcit/Δk and will be used to discriminate changes in ΔUcit/Δk due to filtered load vs renal handling.

CONTACTS AND LOCATIONS:
Overall Officials: Eleanor Lederer, MD, Principal Investigator — University of Texas Southwestern Medical Center

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in this article, after deidentification (text, tables, figures, and appendices) for individual participant data meta-analysis.
Supporting Information: Study Protocol
Time Frame: Beginning 9 months and ending 36 months following article publication.
Access Criteria: Investigators whose proposed use of the data has been approved by an independent review committee ("learned intermediary") identified for this purpose. After 36 months the data will be available in the University's data warehouse but without investigator support other than deposited metadata.